CLINICAL TRIAL: NCT00262002
Title: A Phase II, Randomized, Open Label, Controlled, Multicenter Study to Evaluate the Safety, Immunogenicity and Induction of Immunological Memory After Two or Three Doses of Novartis (Formerly Chiron) Meningococcal ACWY Conjugate Vaccine Administered to Healthy Infants at 2, 3, 4 or 2, 4, 6 Months of Age
Brief Title: Study of the Safety and Immune Response of a Meningococcal Vaccine Administered to Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P5; 2004-000195-13
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Prevention of Meningococcal Disease
MeSH Terms: interventions — Hepatitis B Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; Rubella Vaccine; Tetanus Toxoid

ARMS (7):
- UK234+ (MenACWY Ad+ at 2, 3, 4 m) (Experimental): Three doses of MenACWY Ad+ vaccine were given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age in the UK group. A fourth dose of MenACWY Ad+ was given at 12 months of age.
  Interventions: Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)
- UK24+ (MenACWY Ad+ at 2, 4 m) (Experimental): Two doses of MenACWY Ad+ vaccine were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad+ vaccine was given at 12 months of age.
  Interventions: Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)
- UKMenC (Menjugate at 2, 4 m) (Experimental): Two doses of Menjugate were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. One dose of MenACWY Ad+ vaccine was given at 12 months of age.
  Interventions: Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine); Biological: Menjugate (Men C conjugated vaccine)
- CA246+ (MenACWY Ad+ at 2, 4, 6 m) (Experimental): Three doses of MenACWY Ad+ vaccine were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age of the Canadian group (Prevnar at 6 months was optional and was given if available).One subgroup of subjects was given a reduced dose (1/5) of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
  Interventions: Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation); Biological: MenACWY PS (MenACWY-CRM, polysaccharide vaccine); Biological: HBV (Hepatitis B vaccine); Biological: Prevnar (pneumococcal polysaccharide serotypes 4, 9V, 14, 18C, 19F, 23F & 6B conjugated to the CRM197); Biological: MMR (Measles, Mumps and Rubella vaccine); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)
- CA24+ (MenACWY Ad+ at 2, 4 m) (Experimental): Two doses of MenACWY Ad+ vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad+ vaccine or one reduced dose (1/5) of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
  Interventions: Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation); Biological: MenACWY PS (MenACWY-CRM, polysaccharide vaccine); Biological: HBV (Hepatitis B vaccine); Biological: Prevnar (pneumococcal polysaccharide serotypes 4, 9V, 14, 18C, 19F, 23F & 6B conjugated to the CRM197); Biological: MMR (Measles, Mumps and Rubella vaccine); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)
- UK24- (MenACWY Ad- at 2, 4 m) (Experimental): Two doses of MenACWY Ad- vaccine were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad- vaccine was given at 12 months of age.
  Interventions: Biological: MenACWY Ad- (MenACWY-CRM, non adjuvanted formulation); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)
- CA24- (MenACWY Ad- at 2, 4 m) (Experimental): Two doses of MenACWY Ad- vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
  Interventions: Biological: MenACWY Ad- (MenACWY-CRM, non adjuvanted formulation); Biological: MenACWY PS (MenACWY-CRM, polysaccharide vaccine); Biological: HBV (Hepatitis B vaccine); Biological: Prevnar (pneumococcal polysaccharide serotypes 4, 9V, 14, 18C, 19F, 23F & 6B conjugated to the CRM197); Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine)

INTERVENTIONS:
Biological: MenACWY Ad- (MenACWY-CRM, non adjuvanted formulation) — MenACWY-CRM conjugate vaccine formulated without adjuvant was injected IM (intramuscularly) in the anterolateral area of the right thigh.
  Arms: CA24- (MenACWY Ad- at 2, 4 m); UK24- (MenACWY Ad- at 2, 4 m)
Biological: MenACWY Ad+ (MenACWY-CRM, adjuvanted formulation) — MenACWY-CRM conjugate vaccine formulated with adjuvant was injected IM in the anterolateral area of the right thigh.
  Arms: CA24+ (MenACWY Ad+ at 2, 4 m); CA246+ (MenACWY Ad+ at 2, 4, 6 m); UK234+ (MenACWY Ad+ at 2, 3, 4 m); UK24+ (MenACWY Ad+ at 2, 4 m); UKMenC (Menjugate at 2, 4 m)
Biological: MenACWY PS (MenACWY-CRM, polysaccharide vaccine) — MenACWY polysaccharide vaccine was injected in the anterolateral area of the right thigh.
  Arms: CA24+ (MenACWY Ad+ at 2, 4 m); CA24- (MenACWY Ad- at 2, 4 m); CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Biological: HBV (Hepatitis B vaccine) — Hepatitis B vaccine at 2, 4, 6 months of age administered IM in the anterolateral area of the left thigh.
  Arms: CA24+ (MenACWY Ad+ at 2, 4 m); CA24- (MenACWY Ad- at 2, 4 m); CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Biological: Prevnar (pneumococcal polysaccharide serotypes 4, 9V, 14, 18C, 19F, 23F & 6B conjugated to the CRM197) — Prevnar was administered IM in the anterolateral area of the left thigh.
  Arms: CA24+ (MenACWY Ad+ at 2, 4 m); CA24- (MenACWY Ad- at 2, 4 m); CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Biological: MMR (Measles, Mumps and Rubella vaccine) — MMR at 12 month of age, administered in the left arm.
  Arms: CA24+ (MenACWY Ad+ at 2, 4 m); CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Biological: DTaPHibIPV (Diphtheria, Tetanus, acellular Pertussis, H. Influenzae type b, Inactivated Poliovaccine) — DTaPHibIPV at 2, 3, 4 months of age, administered IM in the anterolateral area of the left thigh.
Biological: Menjugate (Men C conjugated vaccine) — Menjugate was injected IM in the anterolateral area of the right thigh.
  Arms: UKMenC (Menjugate at 2, 4 m)

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and induction of immune memory after two or three doses of Novartis (Formerly Chiron) Meningococcal ACWY Conjugate Vaccine administered to healthy infants.

ELIGIBILITY:
Inclusion Criteria

Individuals eligible for enrollment in this study were male, and female infants:

* Who were healthy 2-month old infants (55-89 days, inclusive) born after full term pregnancy with an estimated gestational age ≥ 37 weeks, and a birth weight ≥ 2.5 kg;
* For whom a parent/legal guardian has given written informed consent after the nature of the study has been explained;
* Who were available for all the visits scheduled in the study;
* Who were in good health as determined by:

  * Medical history;
  * Physical examination;
  * Clinical judgment of the investigator.

Exclusion Criteria

Ineligible for the study were infants:

* Whose parents/legal guardians were unwilling, or unable to give written informed consent for the subject to participate in the study;
* Who previously received any meningococcal vaccine;
* Who received prior vaccination with D, T, P (acellular, or whole cell), IPV, or OPV, HBV, H influenzae type b (Hib), or Pneumococcus;
* Who had a previously ascertained or suspected disease caused by N meningitidis, C diphtheriae, C tetani, Poliovirus, Hepatitis B, Hib, Pneumococcus, or B pertussis (history of laboratory-confirmed or clinical condition of spasmodic cough for a period ≥ 2 weeks associated with apnea or whooping cough);
* Who had household contact with and/or intimate exposure to an individual with laboratory-confirmed N meningitis (serogroups A, C, W-135, or Y), B pertussis, Hib, C diphtheriae, Polio, or pneumococcal infection since birth;
* Who had a history of any anaphylactic shock, asthma, urticaria, or other allergic reaction after previous vaccinations, or known hypersensitivity to any vaccine component;
* Who had experienced significant acute or chronic infection within the previous 7 days, or fever (≥ 38.0°C) within the previous 3 days;
* Who had any present, or suspected serious, acute (e.g., leukemia, lymphomas), or chronic disease (e.g., with signs of cardiac, renal failure, or severe malnutrition, or insulin-dependent diabetes); or progressive neurological disease; or a genetic anomaly or known cytogenic disorders (e.g., Downs syndrome);
* Who had a known or suspected autoimmune disease or impairment /alteration of immune function resulting from (for example):

  * receipt of any immunosuppressive therapy since birth;
  * receipt of immunostimulant since birth;
  * receipt of any systemic corticosteroid since birth.
* Who had a suspected or known HIV infection, or HIV-related disease;
* Who had ever received blood, blood products and/or plasma derivatives, or any parenteral immunoglobulin preparation;
* Who had a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* Who had a history of seizure disorder:

  * Febrile seizure;
  * Any other seizure disorder.
* Who had taken systemic antibiotics (either oral or parenteral) within the previous 14 days (EXCEPTION: subjects who received an oral or parenteral β-lactam antibiotic [examples: penicillin, amoxicillin, ceftriaxone, cefuroxime, cephalexin, etc.] may be enrolled 7 days following the last dose);
* Who with their parents/legal guardians were planning to leave the area of the study site before the end of the study period;
* Who had any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
* Who had taken any antipyretic medication in the previous 6 hours.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 601 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Director — Novartis Vaccines & Diagnostics
Locations (3):
- Canada (2):
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - Clinical Trial Research Center, Halifax, Nova Scotia
- Oxford Vaccine Group, Oxford, United Kingdom

REFERENCES:
- [Result] Snape MD, Perrett KP, Ford KJ, John TM, Pace D, Yu LM, Langley JM, McNeil S, Dull PM, Ceddia F, Anemona A, Halperin SA, Dobson S, Pollard AJ. Immunogenicity of a tetravalent meningococcal glycoconjugate vaccine in infants: a randomized controlled trial. JAMA. 2008 Jan 9;299(2):173-84. doi: 10.1001/jama.2007.29-c. PMID 18182599
- [Result] Perrett KP, Snape MD, Ford KJ, John TM, Yu LM, Langley JM, McNeil S, Dull PM, Ceddia F, Anemona A, Halperin SA, Dobson S, Pollard AJ. Immunogenicity and immune memory of a nonadjuvanted quadrivalent meningococcal glycoconjugate vaccine in infants. Pediatr Infect Dis J. 2009 Mar;28(3):186-93. doi: 10.1097/INF.0b013e31818e037d. PMID 19209097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at two centers in Canada and one in UK.
Pre-assignment Details: The two selected countries provided data on different infant vaccination schedules (at 2 and 4 months of age; at 2, 3, and 4 months of age: and at 2, 4, and 6 months of age), and on different recommended concomitant vaccinations.
Groups:
- UK234+ (MenACWY Ad+ at 2,3,4 m): Three doses of MenACWY Ad+ vaccine were given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age. A fourth dose of MenACWY Ad+ was given at 12 months of age.
- UK24+ (MenACWY Ad+ at 2,4 m): Two doses of MenACWY Ad+ vaccine were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad+ vaccine was given at 12 months of age.
- UKMenC (Menjugate at 2,4m): Two doses of Menjugate were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. One dose of MenACWY Ad+ vaccine was given at 12 months of age.
- CA246+ (MenACWY Ad+ at 2,4,6m): Three doses of MenACWY Ad+ vaccine were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
- CA24+ (MenACWY Ad+ at 2,4m): Two doses of MenACWY Ad+ vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- UK24- (MenACWY Ad- at 2,4m): Two doses of MenACWY Ad- vaccine were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad- vaccine was given at 12 months of age.
- CA24- (MenACWY Ad- at 2,4m): Two doses of MenACWY Ad- vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Period: Overall Study
Arm/Group | UK234+ (MenACWY Ad+ at 2,3,4 m) | UK24+ (MenACWY Ad+ at 2,4 m) | UKMenC (Menjugate at 2,4m) | CA246+ (MenACWY Ad+ at 2,4,6m) | CA24+ (MenACWY Ad+ at 2,4m) | UK24- (MenACWY Ad- at 2,4m) | CA24- (MenACWY Ad- at 2,4m)
Started | 90 | 90 | 45 | 98 | 98 | 90 | 90
Completed | 79 | 84 | 45 | 93 | 91 | 83 | 84
Not Completed | 11 | 6 | 0 | 5 | 7 | 7 | 6
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0 | 1 | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Inapropriate enrollment | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 2 | 0 | 2 | 5 | 3 | 2
Not completed — Unable to classify | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- CA24+ (MenACWY Ad+ at 2,4m): Two doses of MenACWY Ad+ vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- CA24- (MenACWY Ad- at 2,4m): Two doses of MenACWY Ad- vaccine were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- Total: Total of all reporting groups
Arm/Group | UK234+ (MenACWY Ad+ at 2,3,4 m) | UK24+ (MenACWY Ad+ at 2,4 m) | UKMenC (Menjugate at 2,4m) | CA246+ (MenACWY Ad+ at 2,4,6m) | CA24+ (MenACWY Ad+ at 2,4m) | UK24- (MenACWY Ad- at 2,4m) | CA24- (MenACWY Ad- at 2,4m) | Total
Number analyzed (Participants) | 90 | 90 | 45 | 98 | 98 | 90 | 90 | 601
Age, Continuous [Mean (Standard Deviation); unit: days] | 62.1 (5.4) | 61.3 (5.0) | 62.6 (6.5) | 65.6 (6.9) | 65.8 (6.9) | 64.1 (5.5) | 69.4 (10.0) | 64.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 26 | 52 | 49 | 48 | 44 | 304
  Male | 46 | 49 | 19 | 46 | 49 | 42 | 46 | 297

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 Against N. Meningitidis Serogroups A, C, W, and Y Following 3 Doses of MenACWY Ad+ Vaccine
Description: Immunogenicity was measured as the percentage of subjects with human serum bactericidal assay (hSBA) titers ≥ 1:4 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W and Y, at the baseline and 1 month after primary vaccination by groups.
Time Frame: Baseline and at 1 month after the 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- UK234+ (MenACWY Ad+ at 2, 3, 4 m): Three doses of MenACWY conjugate vaccine with adjuvant vaccine were given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age. A fourth dose of MenACWY Ad+ was given at 12 months of age.
- CA246+ (MenACWY Ad+ at 2, 4, 6 m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Number analyzed (Participants) | 81 | 87
percentages of subjects
  Ser A - baseline (n=69,80) | 6 [2 to 14] | 0 [0 to 5]
  Ser A - 1 month after primary vacc (n=69,80) | 93 [84 to 98] | 81 [71 to 89]
  Ser C - baseline (n=79,86) | 18 [10 to 28] | 15 [8 to 24]
  Ser C - 1 month after primary vacc (n=79,86) | 96 [89 to 99] | 98 [92 to 100]
  Ser W - baseline (n=69,78) | 54 [41 to 66] | 31 [21 to 42]
  Ser W - 1 month after primary vacc (n=69,78) | 97 [90 to 100] | 99 [93 to 100]
  Ser Y - baseline | 21 [13 to 31] | 17 [10 to 27]
  Ser Y - 1 month after primary vacc | 94 [86 to 98] | 98 [92 to 100]

2. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 Against N. Meningitidis Serogroups A, C, W, and Y Following 3 Doses of MenACWY Ad+ Conjugate Vaccine
Description: Immunogenicity was measured by percentages of subjects With hSBA titers ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W and Y, at baseline and 1 month after primary vaccination by groups.
Time Frame: Baseline and 1 month after the 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- UK234+ (MenACWY Ad+ at 2, 3, 4 m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age. A fourth dose of MenACWY Ad+ was given at 12 months of age.
- CA246+ (MenACWY Ad+ at 2, 4, 6m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6m)
Number analyzed (Participants) | 81 | 87
percentages of subjects
  Ser A - baseline (n=69,80) | 4 [1 to 12] | 0 [0 to 5]
  Ser A - 1 month after primary vacc (n=69,80) | 88 [78 to 95] | 76 [65 to 85]
  Ser C - baseline (n=79,86) | 9 [4 to 17] | 5 [1 to 11]
  Ser C - 1 month after primary vacc (n=79,86) | 92 [84 to 97] | 98 [92 to 100]
  Ser W - baseline (n=69,78) | 46 [34 to 59] | 28 [19 to 40]
  Ser W - 1 month after primary vacc (n=69,78) | 88 [78 to 95] | 96 [89 to 99]
  Ser Y - baseline | 14 [7 to 23] | 11 [6 to 20]
  Ser Y - 1 month after primary vaccination | 93 [85 to 97] | 89 [80 to 94]

3. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) Following 3 Doses of MenACWY Ad+ Conjugate Vaccine
Description: Immunogenicity was measured as hSBA GMTs and associated 95% CI, against N meningitis serogroups A, C, W, and Y, at the baseline and 1 month after primary vaccination by groups.
Time Frame: Baseline and 1 month after the 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Number analyzed (Participants) | 81 | 87
titers
  Ser A - baseline (n=69,80) | 2.2 [2.04 to 2.38] | 2 [1.86 to 2.15]
  Ser A - 1 month after primary vacc (n=69,80) | 53 [38 to 74] | 21 [15 to 29]
  Ser C - baseline (n=79,86) | 2.79 [2.36 to 3.31] | 2.64 [2.25 to 3.11]
  Ser C - 1 month after primary vacc (n=79,86) | 79 [56 to 112] | 124 [89 to 172]
  Ser W - baseline (n=69,78) | 5.76 [4.39 to 7.57] | 4.03 [3.12 to 5.21]
  Ser W - 1 month after primary vacc (n=69,78) | 65 [46 to 92] | 73 [53 to 102]
  Ser Y - baseline | 2.72 [2.34 to 3.17] | 2.64 [2.28 to 3.05]
  Ser Y - 1 month after primary vacc | 56 [41 to 77] | 2.64 [2.28 to 3.05]

4. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 or ≥ 1:8 Against N. Meningitidis Serogroups A, C, W, and Y Following 2 Doses of Novartis MenACWY Ad+ or Novartis MenACWY Ad- Conjugate Vaccines
Description: Immunogenicity was measured as the percentages of subjects With hSBA titers ≥ 1:4 and ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y, at Baseline and 1 month after second vaccination by groups.
Time Frame: Baseline and 1 month after second vaccination
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- UK24+ (MenACWY Ad+ at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad+ vaccine was given at 12 months of age.
- CA24+ (MenACWY Ad+ at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad+ vaccine or one reduced dose (one fifth) of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- UK24- (MenACWY Ad- at 2, 4 m): Two doses of MenACWY conjugate vaccine without adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad- vaccine was given at 12 months of age.
- CA24- (MenACWY Ad- at 2, 4 m): Two doses of MenACWY conjugate vaccine without adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age. One dose of MenACWY Ad- vaccine or one reduced dose (one fifth) of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK24+ (MenACWY Ad+ at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 77 | 79 | 79 | 85
percentages of subjects
  Ser A - hSBA ≥1:4, baseline (N=68,79,78,83) | 4 [1 to 12] | 3 [0 to 9] | 3 [0 to 9] | 4 [1 to 10]
  Ser A - hSBA ≥1:4, 1m after 2n vacc(N=68,79,78,83) | 60 [48 to 72] | 66 [54 to 76] | 50 [38 to 62] | 57 [45 to 67]
  Ser A - hSBA ≥1:8, baseline (N=68,79,78,83) | 3 [0 to 10] | 1 [0.032 to 7] | 0 [0 to 5] | 1 [0.03 to 7]
  Ser A - hSBA≥1:8, 1m after 2nd vacc(N=68,79,78,83) | 54 [42 to 67] | 58 [47 to 69] | 44 [32 to 55] | 49 [38 to 61]
  Ser C - hSBA ≥1:4, baseline (N=77,74,79,85) | 13 [6 to 23] | 15 [8 to 25] | 20 [12 to 31] | 20 [12 to 30]
  Ser C - hSBA ≥1:4,1m after 2nd vacc(N=77,74,79,85) | 84 [74 to 92] | 91 [81 to 96] | 86 [76 to 93] | 93 [85 to 97]
  Ser C - hSBA ≥1:8, baseline (N=77,74,79,85) | 9 [4 to 18] | 15 [8 to 25] | 5 [1 to 12] | 11 [5 to 19]
  Ser C - hSBA ≥1:8,1m after 2nd vacc(N=77,74,79,85) | 83 [73 to 91] | 85 [75 to 92] | 82 [72 to 90] | 89 [81 to 95]
  Ser W - hSBA ≥1:4, baseline (N=73,74,72,75) | 45 [34 to 57] | 24 [15 to 36] | 43 [31 to 55] | 19 [11 to 29]
  Ser W - hSBA ≥1:4,1m after 2nd vacc(N=73,74,72,75) | 92 [83 to 97] | 91 [81 to 96] | 82 [71 to 90] | 95 [87 to 99]
  Ser W - hSBA ≥1:8, baseline (N=73,74,72,75) | 37 [26 to 49] | 19 [11 to 30] | 36 [25 to 48] | 16 [9 to 26]
  Ser W -hSBA ≥1:8,1m after 2nd vacc(N=73,74,72,75) | 84 [73 to 91] | 85 [75 to 92] | 75 [63 to 84] | 92 [83 to 97]
  Ser Y - hSBA ≥1:4, baseline (N=76,74,77,85) | 18 [10 to 29] | 9 [4 to 19] | 35 [25 to 47] | 18 [10 to 27]
  Ser Y -hSBA ≥1:4,1m after 2nd vacc(N=76,74,77,85) | 84 [74 to 92] | 86 [77 to 93] | 74 [63 to 83] | 91 [82 to 96]
  Ser Y - hSBA ≥1:8, baseline (N=76,74,77,85) | 7 [2 to 15] | 4 [1 to 11] | 16 [8 to 26] | 11 [5 to 19]
  Ser Y -hSBA ≥1:8,1m after 2nd vacc(N=76,74,77,85) | 76 [65 to 85] | 80 [69 to 88] | 70 [59 to 80] | 86 [77 to 92]

5. Secondary Outcome: Geometric Mean hSBA Titer (GMTs) Following 2 Doses of MenACWY Ad+ and MenACWY Ad- Conjugate Vaccines
Description: Immunogenicity was measured as hSBA GMTs and associated 95% CI against N. Meningitidis serogroups A, C, W, and Y at baseline and 1 month after second vaccination by groups.
Time Frame: Baseline and 1 month after second vaccination
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- CA24+ (MenACWY Ad+ at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age. One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- CA24- (MenACWY Ad- at 2, 4 m): Two doses of MenACWY conjugate vaccine without adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age. One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK24+ (MenACWY Ad+ at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 77 | 79 | 79 | 85
titers
  Ser A - baseline (n=68,79,78,83) | 2.17 [2.01 to 2.35] | 2.07 [1.93 to 2.23] | 2.05 [1.91 to 2.21] | 2.08 [1.94 to 2.23]
  Ser A - 1 month after 2nd vacc (n=68,79,78,83) | 12 [8.36 to 16] | 11 [7.91 to 15] | 7.3 [5.31 to 10] | 7.16 [5.26 to 9.73]
  Ser C - baseline (n=77,74,79,85) | 2.54 [2.14 to 3.02] | 2.77 [2.33 to 3.31] | 2.48 [2.09 to 2.94] | 2.87 [2.44 to 3.39]
  Ser C - 1 month after 2nd vacc (n=77,74,79,85) | 52 [37 to 74] | 55 [38 to 79] | 40 [28 to 57] | 69 [49 to 96]
  Ser W - baseline (n=73,74,79,75) | 5.33 [4.09 to 6.94] | 3.6 [2.77 to 4.69] | 5.14 [3.94 to 6.71] | 3.02 [2.33 to 3.93]
  Ser W - 1 month after 2nd vacc (n=73,74,79,75) | 48 [34 to 67] | 44 [31 to 61] | 29 [20 to 40] | 69 [50 to 96]
  Ser Y - baseline (n=76,74,77,85) | 2.56 [2.19 to 2.99] | 2.27 [1.94 to 2.66] | 3.39 [2.9 to 3.96] | 2.76 [2.38 to 3.21]
  Ser Y - 1 month after 2nd vacc (n=76,74,77,85) | 26 [19 to 37] | 27 [19 to 38] | 21 [15 to 29] | 41 [30 to 56]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 or ≥ 1:8 Against N. Meningitidis Serogroups A, C, W & Y After a Booster Dose of MenACWY Ad+ or Ad- Vaccine in a Subgroup of Subjects Following 2 or 3 Doses or MenACWY Ad+ or 2 Doses of MenACWY Ad- Vaccine
Description: Immunogenicity was measured as the percentages of subjects with hSBA ≥ 1:4 or ≥ 1:8 and associated 95% CI, against N. Meningitidis serogroups A, C, W, and Y, at 12 months of age and 1 month after booster by groups.
Time Frame: at 12 months of age and 1 month after booster vaccination
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | UK24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 67 | 63 | 65 | 40 | 40
percentages of subjects
  Ser A -hSBA ≥1:4, at 12 m of age(n=64,61,62,39,38) | 8 [3 to 17] | 7 [2 to 16] | 21 [12 to 33] | 5 [1 to 17] | 3 [0.067 to 14]
  Ser A -hSBA≥1:4, 1 m after booster vacc | 86 [75 to 93] | 79 [66 to 88] | 94 [84 to 98] | 92 [79 to 98] | 95 [82 to 99]
  Ser A - hSBA ≥1:8, at 12 months of age | 5 [1 to 13] | 5 [1 to 14] | 13 [6 to 24] | 3 [0.065 to 13] | 3 [0.067 to 14]
  Ser A - hSBA ≥1:8, 1 m after booster vaccination | 83 [71 to 91] | 77 [65 to 87] | 92 [82 to 97] | 90 [76 to 97] | 92 [79 to 98]
  Ser C -hSBA ≥1:4, at 12 m of age(n=67,63,65,40,40) | 40 [28 to 53] | 33 [22 to 46] | 60 [47 to 72] | 48 [32 to 64] | 33 [19 to 49]
  Ser C-hSBA≥1:4,1 m after booster(n=57,63,65,40,40) | 96 [87 to 99] | 94 [85 to 98] | 98 [92 to 100] | 98 [87 to 100] | 100 [91 to 100]
  Ser C-hSBA ≥1:8, at 12 m of age(n=67,40,65,40,40) | 34 [23 to 47] | 27 [17 to 40] | 52 [40 to 65] | 35 [21 to 52] | 25 [13 to 41]
  Ser C-hSBA≥1:8, 1m after booster(n=67,63,65,40,40) | 96 [87 to 99] | 94 [85 to 98] | 98 [92 to 100] | 95 [83 to 99] | 100 [91 to 100]
  Ser W -hSBA≥1:4, at 12 m of age(n=57,41,57,35,35) | 56 [42 to 69] | 54 [37 to 69] | 81 [68 to 90] | 74 [57 to 88] | 69 [51 to 83]
  Ser W - hSBA≥1:4, 1m after booster vaccination | 100 [94 to 100] | 100 [91 to 100] | 100 [94 to 100] | 100 [90 to 100] | 100 [90 to 100]
  Ser W -hSBA≥1:8, at 12 m of age(n=57,41,40,35,35) | 47 [34 to 61] | 41 [26 to 58] | 68 [55 to 80] | 49 [31 to 66] | 54 [37 to 71]
  Ser W -hSBA≥1:8,1m after booster(n=57,41,57,35,35) | 100 [94 to 100] | 100 [91 to 100] | 100 [94 to 100] | 100 [90 to 100] | 100 [90 to 100]
  Ser Y -hSBA≥1:4, at 12m of age(n=66,63,65,40,38) | 52 [39 to 64] | 52 [39 to 65] | 86 [75 to 93] | 65 [48 to 79] | 63 [46 to 78]
  Ser Y - hSBA≥1:4, 1 m after booster vaccination | 100 [95 to 100] | 100 [94 to 100] | 100 [94 to 100] | 100 [91 to 100] | 100 [91 to 100]
  Ser Y - hSBA ≥1:8, at 12 months of age | 39 [28 to 52] | 41 [29 to 54] | 72 [60 to 83] | 45 [29 to 62] | 53 [36 to 69]
  Ser Y - hSBA ≥1:8, 1 m after booster vaccination | 100 [95 to 100] | 100 [94 to 100] | 100 [94 to 100] | 100 [91 to 100] | 100 [91 to 100]

7. Secondary Outcome: Geometric Mean hSBA Titers (GMT) After a Booster Dose of MenACWY Ad+ or Ad- Vaccine Conjugate in a Subgroup of Subjects Following Either 2 or 3 Doses of MenACWY Ad+ Vaccine or 2 Doses of MenACWY Ad- Conjugate Vaccines
Description: Immunogenicity was measured as GMT and associated 95% CI against N. Meningitidis serogroups A, C, W, and Y, at 12 months of age and 1 month after booster by group.
Time Frame: at 12 months of age and 1 month after booster vaccination
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- CA24+ (MenACWY Ad+ at 2, 4m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA24+ (MenACWY Ad+ at 2, 4m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 67 | 63 | 65 | 40 | 40
titers
  Ser A - at 12 months of age (n=64,61,62,39,38) | 2.31 [2 to 2.66] | 2.22 [1.92 to 2.57] | 2.97 [2.57 to 3.44] | 2.18 [1.74 to 2.73] | 2.07 [1.65 to 2.6]
  Ser A - 1 month after booster (n=64,61,62,39,38) | 47 [31 to 72] | 30 [19 to 47] | 134 [87 to 207] | 67 [43 to 106] | 59 [38 to 93]
  Ser C - at 12 months of age(n=67,63,65,40,40) | 5.18 [3.83 to 7.02] | 3.94 [2.88 to 5.39] | 7.94 [5.84 to 11] | 4.64 [3.11 to 6.91] | 4.07 [2.73 to 6.06]
  Ser C - 1 month after booster(n=67,63,65,40,40) | 236 [159 to 349] | 129 [86 to 194] | 429 [288 to 639] | 216 [130 to 356] | 258 [56 to 426]
  Ser W - at 12 months of age(n=57,41,57,35,35) | 8.1 [5.76 to 11] | 6.49 [4.34 to 9.7] | 16 [11 to 23] | 8.84 [5.63 to 14] | 11 [7.04 to 17]
  Ser W - 1 month after booster (n=57,41,57,35,35) | 503 [347 to 732] | 311 [200 to 485] | 792 [544 to 1154] | 381 [224 to 650] | 402 [236 to 684]
  Ser Y - at 12 months of age (n=66,63,65,40,38) | 6.65 [4.88 to 9.06] | 6.83 [4.98 to 9.37] | 19 [14 to 26] | 7.99 [5.29 to 12] | 7.63 [5 to 12]
  Ser Y- 1 month after booster(n=66,63,65,40,38) | 508 [358 to 723] | 438 [305 to 628] | 1395 [979 to 1989] | 308 [191 to 499] | 527 [322 to 862]

8. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 and ≥ 1:8 Against N. Meningitidis Serogroups A, C, W and Y Following 2 Doses of Novartis MenACWY Ad+ Vaccine, Novartis MenACWY Ad- Vaccine or Novartis Menjugate Vaccine
Description: The persistence of immune response was measured as the percentages of subjects with hSBA ≥ 1:4 and ≥ 1:8 against N. Meningitidis serogroups A, C, W, and Y at 12 months of age by groups.
Time Frame: at 12 months of age
Population: The analysis was performed on the MenACWY and Menjugate per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- UKMenC (Menjugate 2, 4 m): Two doses of Menjugate were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. One dose of MenACWY Ad+ vaccine was given at 12 months of age.
- CA24+ (MenACWY Ad+ at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad+ vaccine or one reduced dose ( of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UKMenC (Menjugate 2, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 38 | 69 | 66 | 77 | 81
percentages of subjects
  Ser A - hSBA ≥1:4, at 12m of age(n=36,62,65,77,78) | 0 [0 to 10] | 8 [3 to 18] | 6 [2 to 15] | 8 [3 to 16] | 5 [1 to 13]
  Ser A - hSBA ≥1:8, at 12m of age(n=36,62,65,77,78) | 0 [0 to 10] | 5 [1 to 13] | 5 [1 to 13] | 5 [1 to 13] | 4 [1 to 11]
  Ser C - hSBA ≥1:4, at 12m of age(n=38,69,69,73,81) | 89 [75 to 97] | 41 [29 to 53] | 32 [21 to 44] | 48 [36 to 60] | 35 [24 to 46]
  Ser C - hSBA ≥1:8, at 12m of age(n=38,69,69,73,81) | 87 [72 to 96] | 33 [22 to 46] | 26 [16 to 38] | 40 [28 to 52] | 30 [20 to 41]
  Ser W - hSBA ≥1:4, at 12m of age(n=34,62,42,69,69) | 9 [2 to 24] | 58 [45 to 70] | 57 [41 to 72] | 64 [51 to 75] | 75 [64 to 85]
  Ser W - hSBA ≥1:8, at 12m of age(n=34,62,42,69,69) | 6 [1 to 20] | 48 [35 to 61] | 45 [30 to 61] | 52 [40 to 64] | 61 [48 to 72]
  Ser Y - hSBA ≥1:4, at 12m of age(n=38,69,66,73,79) | 5 [1 to 18] | 51 [38 to 63] | 56 [43 to 68] | 60 [48 to 72] | 59 [48 to 70]
  Ser Y - hSBA ≥1:8, at 12m of age(n=38,69,66,73,79) | 3 [0.067 to 14] | 42 [30 to 55] | 45 [33 to 58] | 51 [39 to 63] | 46 [34 to 57]

9. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) After 2 Doses of Novartis MenACWY Ad+ Vaccines, Novartis MenACWY Ad- Vaccine, or Novartis Menjugate Vaccine.
Description: The persistence of immune response as measured by hSBA GMT and associated 95% CI against N. Meningitidis serogroups A, C, W, and Y, at 12 months of age by groups.
Time Frame: at 12 months of age
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | UKMenC (Menjugate at 2, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 38 | 69 | 66 | 77 | 81
titers
  Ser A - at 12 months of age (n=36,62,65,77,78) | 2 [1.62 to 2.48] | 2.32 [1.97 to 2.73] | 2.2 [1.88 to 2.58] | 2.29 [1.98 to 2.65] | 2.18 [1.89 to 2.52]
  Ser C - at 12 months of age (n=36,69,69,73,82) | 27 [18 to 40] | 5.04 [3.73 to 6.81] | 3.85 [2.85 to 5.21] | 5.43 [4.05 to 7.27] | 4.42 [3.35 to 5.84]
  Ser W - at 12 months of age (n=34,62,42,69,69) | 2.42 [1.55 to 3.78] | 8.38 [6.03 to 12] | 7.02 [4.71 to 10] | 8.15 [5.97 to 11] | 12 [8.81 to 16]
  Ser Y - at 12 months of age (n=38,69,66,73,79) | 2.15 [1.41 to 3.28] | 6.72 [4.92 to 9.18] | 7.64 [5.55 to 11] | 7.84 [5.79 to 11] | 7.12 [5.32 to 9.54]

10. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 and ≥ 1:8 Against N. Meningitidis Serogroup A, C, W and Y Following 3 Doses of Novartis MenACWY Ad+ Conjugate Vaccine
Description: The persistence of immune response as measured by percentages of subjects with hSBA≥ 1:4 and hSBA ≥ 1:8 and associated 95% CI, against N. Meningitidis serogroups A, C, W, and Y, at 12 months by groups.
Time Frame: at 12 months of age
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Number analyzed (Participants) | 71 | 86
percentages of subjects
  Ser A - hSBA ≥1:4, at 12 months of age (n=58,79) | 21 [11 to 33] | 35 [25 to 47]
  Ser A - hSBA ≥1:8, at 12 months of age(n=58,79) | 16 [7 to 27] | 29 [19 to 40]
  Ser C - hSBA ≥1:4, at 12 months of age(n=70,84) | 59 [46 to 70] | 75 [64 to 84]
  Ser C - hSBA ≥1:8, at 12 months of age(n=70,84) | 47 [35 to 59] | 68 [57 to 78]
  Ser W - hSBA ≥1:4, at 12 months of age(n=58,75) | 78 [65 to 87] | 89 [80 to 95]
  Ser W - hSBA ≥1:8, at 12 months of age(n=58,75) | 66 [52 to 78] | 81 [71 to 89]
  Ser Y - hSBA ≥1:4, at 12 months of age(n=71,86) | 85 [74 to 92] | 87 [78 to 93]
  Ser Y - hSBA ≥1:8, at 12 months of age(n=71,86) | 70 [58 to 81] | 79 [69 to 87]

11. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) Following 3 Doses of Novartis MenACWY Ad+ Conjugate Vaccine
Description: The persistence of immune response as measured by hSBA GMTs and associated 95% CI against N. Meningitidis serogroups A, C, W, and Y,at 12 months by groups.
Time Frame: at 12 months of age
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Number analyzed (Participants) | 71 | 86
Titers
  Ser A - at 12 months of age (n=58,79) | 3.02 [2.55 to 3.57] | 3.93 [3.4 to 4.54]
  Ser C - at 12 months of age (n=70,84) | 7.56 [5.61 to 10] | 14 [10 to 18]
  Ser W - at 12 months of age (n=58,75) | 15 [10 to 21] | 20 [15 to 27]
  Ser Y - at 12 months of age (n=71,86) | 18 [13 to 24] | 22 [17 to 29]

12. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 or ≥ 1:8 in Subjects Challenged With a Reduced Dose of Licensed Meningococcal ACWY PS Vaccine Following 3 Doses of Novartis MenACWY Ad+ Conjugate Vaccine
Description: The induction of immunological memory was measured as percentages of subjects with hSBA ≥ 1:4 and hSBA ≥ 1:8 and associated 95% CI, against N. Meningitidis serogroups A, C, W, and Y , before challenge at 12 months of age and 1 month after PS challenge.
Time Frame: before challenge at 12 months of age and 1 month after PS challenge.
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- CA246+ (MenACWY Ad+ at 2,4,6 m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | CA246+ (MenACWY Ad+ at 2,4,6 m)
Number analyzed (Participants) | 44
percentages of subjects
  Ser A-hSBA≥1:4,before challenge at 12m (n=44) | 27 [15 to 43]
  Ser A - hSBA ≥1:4, 1 month after PS (n=44) | 89 [75 to 96]
  Ser A-hSBA ≥1:8,before challenge at 12m (n=44) | 23 [11 to 38]
  Ser A - hSBA ≥1:8, 1 month after PS (n=44) | 86 [73 to 95]
  Ser C-hSBA ≥1:4,before challenge at 12m (n=43) | 74 [59 to 86]
  Ser C - hSBA ≥1:4, 1 month after PS (n=43) | 95 [84 to 99]
  Ser C-hSBA ≥1:8, before challenge at 12m (n=43) | 65 [49 to 79]
  Ser C - hSBA ≥1:8, 1 month after PS (n=43) | 91 [78 to 97]
  Ser W-hSBA ≥1:4,before challenge at 12m (n=40) | 83 [67 to 93]
  Ser W - hSBA ≥1:4, 1 month after PS (n=40) | 98 [87 to 100]
  Ser W-hSBA ≥1:8,before challenge at 12m (n=40) | 73 [56 to 85]
  Ser W - hSBA ≥1:8, 1 month after PS (n=40) | 95 [83 to 99]
  Ser Y-hSBA ≥1:4,before challenge at 12m (n=44) | 89 [75 to 96]
  Ser Y - hSBA ≥1:4, 1 month after PS (n=44) | 98 [88 to 100]
  Ser Y-hSBA ≥1:8,before challenge at 12m (N=44) | 77 [62 to 89]
  Ser Y - hSBA ≥1:8, 1 month after PS (n=44) | 98 [88 to 100]

13. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) in Subjects Challenged With a Reduced Dose of Licensed Meningococcal ACWY PS Vaccine Following 3 Doses of Novartis MenACWY Ad+ Conjugate Vaccine
Description: The induction of immunological memory was measured as hSBA Geometric Mean Titers (GMTs) and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y , before challenge at 12 months of age and 1 month after PS challenge.
Time Frame: before challenge at 12 months of age and 1 month after PS challenge.
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- CA246+ (MenACWY Ad+ at 2, 4,6 m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | CA246+ (MenACWY Ad+ at 2, 4,6 m)
Number analyzed (Participants) | 44
titers
  Ser A - before challenge at 12 months of age(n=44) | 3.4 [2.75 to 4.2]
  Ser A - 1 month after PS challenge (n=44) | 32 [21 to 48]
  Ser C - before challenge at 12 months of age(n=43) | 12 [8.41 to 18]
  Ser C - 1 month after PS challenge (n=43) | 82 [50 to 133]
  Ser W - before challenge at 12 months of age(n=40) | 17 [11 to 25]
  Ser W - 1 month after PS challenge (n=40) | 249 [152 to 410]
  Ser Y - before challenge at 12 months of age(n=44) | 19 [13 to 28]
  Ser Y - 1 month after PS challenge (n=44) | 186 [117 to 294]

14. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 or ≥ 1:8 in Subjects Challenged With a Reduced Dose of Licensed Meningococcal ACWY PS Vaccine Following Two Doses of Novartis MenACWY Ad+ or MenACWY Ad- Conjugate Vaccine
Description: The Induction of immunological memory was measured as percentage of subjects with hSBA ≥ 1:4, hSBA ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y, before challenge at 12 months and 1 month after PS challenge by groups.
Time Frame: Before challenge at 12 months of age and 1 month after PS challenge.
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- CA24- (MenACWY Ad- at 2, 4m): Two doses of MenACWY conjugate vaccine without adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | CA24+ (MenACWY Ad+ at 2, 4m) | CA24- (MenACWY Ad- at 2, 4m)
Number analyzed (Participants) | 42 | 39
percentages of subjects
  Ser A - hSBA≥1:4,before challange at 12m (n=40,39) | 8 [2 to 20] | 8 [2 to 21]
  Ser A - hSBA ≥1:4,1 month after PS (n=40,39) | 78 [62 to 89] | 92 [79 to 98]
  Ser A - hSBA≥1:8,before challange at 12m (n=40,39) | 5 [1 to 17] | 5 [1 to 17]
  Ser A - hSBA ≥1:8, 1 month after PS (n=40,39) | 78 [62 to 89] | 87 [73 to 96]
  Ser C - hSBA≥1:4,before challange at 12m (n=41,39) | 44 [28 to 60] | 38 [23 to 55]
  Ser C - hSBA ≥1:4, 1 month after PS (n=41,39) | 95 [83 to 99] | 95 [83 to 99]
  Ser C - hSBA≥1:8,before challange at 12m(n=41,39) | 39 [24 to 55] | 36 [21 to 53]
  Ser C - hSBA ≥1:8, 1 month after PS (n=41,39) | 93 [80 to 98] | 90 [76 to 97]
  Ser W - hSBA ≥1:4,before challange at 12m(n=41,38) | 59 [42 to 74] | 71 [54 to 85]
  Ser W - hSBA ≥1:4, 1 month after PS (n=41,38) | 98 [87 to 100] | 100 [91 to 100]
  Ser W - hSBA ≥1:8,before challange at 12m(n=41,38) | 51 [35 to 67] | 58 [41 to 74]
  Ser W - hSBA ≥1:8, 1 month after PS (n=41,38) | 98 [87 to 100] | 100 [91 to 100]
  Ser Y - hSBA ≥1:4,before challange at 12m(n=42,38) | 55 [39 to 70] | 55 [38 to 71]
  Ser Y - hSBA ≥1:4, 1 month after PS (n=42,38) | 98 [87 to 100] | 100 [91 to 100]
  Ser Y - hSBA ≥1:8,before challange at 12m (n=42,38 | 50 [34 to 66] | 42 [26 to 59]
  Ser Y - hSBA ≥1:8, 1 month after PS (n=42,38) | 98 [87 to 100] | 97 [86 to 100]

15. Secondary Outcome: Geometric Mean hSBA Titers (GMTs) in Subjects Challenged With a Reduced Dose of Licensed Meningococcal ACWY PS Vaccine Following Two Doses of Novartis MenACWY Ad+ or MenACWY Ad- Conjugate Vaccine
Description: Induction of immunological memory was measured by hSBA Geometric Mean Titers (GMTs) and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y, before challenge at 12 months and 1 month after PS challenge by groups.
Time Frame: Before challenge at 12 months of age and 1 month after PS challenge.
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- CA24+ (MenACWY Ad+ at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- CA24- (MenACWY Ad- at 2, 4 m): Two doses of MenACWY conjugate vaccine without adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | CA24+ (MenACWY Ad+ at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 42 | 39
titers
  Ser A - before challenge at 12 months (n=40,39) | 2.22 [1.77 to 2.76] | 2.31 [1.84 to 2.89]
  Ser A - 1 month after PS challenge (n=40,39) | 28 [18 to 44] | 55 [35 to 86]
  Ser C - before challenge at 12 months (n=41,39) | 5.21 [3.51 to 7.72] | 5.07 [3.38 to 7.59]
  Ser C - 1 month after PS challenge (n=41,39) | 140 [85 to 231] | 181 [109 to 301]
  Ser W - before challenge at 12 months (n=41,38) | 7.48 [4.94 to 11] | 11 [7.08 to 17]
  Ser W - 1 month after PS challenge (n=41,38) | 365 [224 to 597] | 555 [333 to 924]
  Ser Y - before challenge at 12 months (n=42,38) | 6.73 [4.51 to 10] | 6.79 [4.45 to 10]
  Ser Y - 1 month after PS challenge (n=42,38) | 280 [175 to 448] | 288 [176 to 472]

16. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:4 and ≥ 1:8 of MenACWY Ad+ Conjugate Vaccine
Description: The immunogenicity was measured as percentages of subject with hSBA≥ 1:4 and hSBA ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y, baseline and 1 month after 2 or 3 dose primary series by groups.
Time Frame: Baseline and 1 month after the 2 or 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- CA246+ (MenACWY Ad+ at 2, 4, 6m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was to be given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6m) | UK24+ (MenACWY Ad+ at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4m)
Number analyzed (Participants) | 81 | 87 | 77 | 79
percentages of subjects
  Ser A - hSBA ≥1:4, baseline (n=69,80,38,79) | 6 [2 to 14] | 0 [0 to 5] | 4 [1 to 12] | 3 [0 to 9]
  Ser A - hSBA≥1:4,1m after 1st vacc (n=69,80,38,79) | 93 [84 to 98] | 81 [71 to 89] | 60 [48 to 72] | 66 [54 to 76]
  Ser A - hSBA ≥1:8, baseline (n=69,80,38,79) | 4 [1 to 12] | 0 [0 to 5] | 3 [0 to 10] | 1 [0.032 to 7]
  Ser A - hSBA≥1:8,1m after 1st vacc (n=69,80,38,79) | 88 [78 to 95] | 76 [65 to 85] | 54 [42 to 67] | 58 [47 to 69]
  Ser C - hSBA ≥1:4, baseline (n=79,86,40,74) | 18 [10 to 28] | 15 [8 to 24] | 13 [6 to 23] | 15 [8 to 25]
  Ser C - hSBA≥1:4,1m after 1st vacc (n=79,86,40,74) | 96 [89 to 99] | 98 [92 to 100] | 84 [74 to 92] | 91 [81 to 96]
  Ser C - hSBA ≥1:8, baseline (n=79,86,40,74) | 9 [4 to 17] | 5 [1 to 11] | 9 [4 to 18] | 15 [8 to 25]
  Ser C - hSBA≥1:8,1m after 1st vacc (n=79,86,40,74) | 92 [84 to 97] | 98 [92 to 100] | 83 [73 to 91] | 85 [75 to 92]
  Ser W - hSBA ≥1:4, baseline (n=69,78,73,74) | 54 [41 to 66] | 31 [21 to 42] | 45 [34 to 57] | 24 [15 to 36]
  Ser W - hSBA≥1:4,1m after 1st vacc (n=69,78,73,74) | 97 [90 to 100] | 99 [93 to 100] | 92 [83 to 97] | 91 [81 to 96]
  Ser W - hSBA ≥1:8, baseline (n=69,78,73,74) | 46 [34 to 59] | 28 [19 to 40] | 37 [26 to 49] | 19 [11 to 30]
  Ser W - hSBA≥1:8,1m after 1st vacc (n=69,78,73,74) | 88 [78 to 95] | 96 [89 to 99] | 84 [73 to 91] | 85 [75 to 92]
  Ser Y - hSBA ≥1:4, baseline (n=81,87,76,74) | 21 [13 to 31] | 17 [10 to 27] | 18 [10 to 29] | 9 [4 to 19]
  Ser Y - hSBA≥1:4,1m after 1st vacc (n=81,87,76,74) | 94 [86 to 98] | 98 [92 to 100] | 84 [74 to 92] | 86 [77 to 93]
  Ser Y - hSBA ≥1:8, baseline (n=81,87,76,74) | 14 [7 to 23] | 11 [6 to 20] | 7 [2 to 15] | 4 [1 to 11]
  Ser Y - hSBA≥1:8,1m after 1st vacc (n=81,87,76,74) | 93 [85 to 97] | 89 [80 to 94] | 76 [65 to 85] | 80 [69 to 88]

17. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:4 and ≥ 1:8 in Subjects Challenged With a Reduced Dose of a Licensed Meningococcal ACWY PS Vaccine Following 2 or 3 Doses of MenACWY Ad+ Conjugate Vaccine
Description: The memory response was measured as percentages of subjects with hSBA ≥ 1:4 and hSBA ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroups A, C, W, and Y, at 12 months of age and 1 month after PS challenge by groups.
Time Frame: at 12 months of age and 1 month after PS challenge
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population evaluating the persistence response.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | CA246+ (MenACWY Ad+ at 2, 4, 6m) | CA24+ (MenACWY Ad+ at 2, 4 m)
Number analyzed (Participants) | 44 | 42
percentages of subjects
  Ser A - hSBA ≥1:4, at 12 months of age (n=44,40) | 27 [15 to 43] | 8 [2 to 20]
  Ser A - hSBA ≥1:4, at 1 month after PS (n=44,40) | 89 [75 to 96] | 78 [62 to 89]
  Ser A - hSBA ≥1:8, at 12 months of age (n=44,40) | 23 [11 to 38] | 5 [1 to 17]
  Ser A - hSBA ≥1:8, at 1 month after PS (n=44,40) | 86 [73 to 95] | 78 [62 to 89]
  Ser C - hSBA ≥1:4, at 12 months of age (n=43,41) | 74 [59 to 86] | 44 [28 to 60]
  Ser C - hSBA ≥1:4, at 1 month after PS (n=43,41) | 95 [84 to 99] | 95 [83 to 99]
  Ser C - hSBA ≥1:8, at 12 months of age (n=43,41) | 65 [49 to 79] | 39 [24 to 55]
  Ser C - hSBA ≥1:8, at 1 month after PS (n=43,41) | 91 [78 to 97] | 93 [80 to 98]
  Ser W - hSBA ≥1:4, at 12 months of age (n=40,41) | 83 [67 to 93] | 59 [42 to 74]
  Ser W - hSBA ≥1:4, at 1 month after PS (n=40,41) | 98 [87 to 100] | 98 [87 to 100]
  Ser W - hSBA ≥1:8, at 12 months of age (n=40,41) | 73 [56 to 85] | 51 [35 to 67]
  Ser W - hSBA ≥1:8, at 1 month after PS (n=40,41) | 95 [83 to 99] | 98 [87 to 100]
  Ser Y - hSBA ≥1:4, at 12 months of age (n=44,42) | 89 [75 to 96] | 55 [39 to 70]
  Ser Y - hSBA ≥1:4, at 1 month after PS (n=44,42) | 98 [88 to 100] | 98 [87 to 100]
  Ser Y - hSBA ≥1:8, at 12 months of age (n=44,42) | 77 [62 to 89] | 50 [34 to 66]
  Ser Y - hSBA ≥1:8, at 1 month after PS (n=44,42) | 98 [88 to 100] | 98 [87 to 100]

18. Secondary Outcome: Percentages of Subjects With Antibody Response to Routine Vaccines (Hib, Diphtheria, Tetanus, Hepatitis B) When Routine Vaccines Are Given Concomitantly With Novartis MenACWY Ad+ or Novartis MenACWY Ad- Conjugate Vaccines
Description: To assess the immunogenicity of routine vaccines when given concomitantly to Novartis MenACWY Ad+ or Novartis MenACWY Ad- conjugate vaccines. Hib, diphtheria, tetanus, pertussis will be evaluated as the first priority, followed by pneumococcus, polio, hepatitis B, and MMR (measles, mumps, and rubella) depending on the availability of sera.
Time Frame: Baseline and 1 month after the 2 or 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m) | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m)
Number analyzed (Participants) | 70 | 77 | 70 | 73 | 72 | 73
percentages of subjects
  Antitetanus≥0.1 IU/mL-baseline(69,71,70,67,69,72) | 75 [64 to 85] | 79 [68 to 88] | 70 [58 to 80] | 93 [83 to 98] | 87 [77 to 94] | 71 [59 to 81]
  Antitetanus≥0.1 IU/mL -1m post (69,71,70,67,69,72) | 100 [95 to 100] | 100 [95 to 100] | 99 [92 to 100] | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100]
  antidipht≥0.1 IU/mL-baseline(69,71,70,67,69,72) | 17 [9 to 28] | 14 [7 to 24] | 3 [0 to 10] | 18 [10 to 29] | 19 [10 to 30] | 15 [8 to 26]
  antidipht≥0.1 IU/mL- 1m post (69,71,70,67,69,72) | 96 [88 to 99] | 97 [90 to 100] | 100 [95 to 100] | 97 [90 to 100] | 96 [88 to 99] | 100 [95 to 100]
  antiPRPtiter≥0.15µg/mL-baseline(70,77,69,73,72,73) | 36 [25 to 48] | 42 [30 to 53] | 17 [9 to 28] | 25 [15 to 36] | 49 [37 to 61] | 37 [26 to 49]
  antiPRPtiter≥0.15µg/mL-1m post (70,77,69,73,72,73) | 74 [62 to 84] | 95 [87 to 99] | 67 [54 to 78] | 97 [90 to 100] | 97 [90 to 100] | 100 [95 to 100]
  antiPRPtiter≥1.0 µg/mL-baseline(70,77,69,73,72,73) | 10 [4 to 20] | 17 [9 to 27] | 3 [0 to 10] | 7 [2 to 15] | 17 [9 to 27] | 11 [5 to 20]
  antiPRPtiter≥1.0 µg/mL-1m post (70,77,69,73,72,73) | 33 [22 to 45] | 86 [76 to 93] | 35 [24 to 47] | 82 [71 to 90] | 82 [71 to 90] | 86 [76 to 93]
  antiHBVtiter≥1.0 IU/mL-baseline(65,na,66,na,na,67) | 23 [14 to 35] | NA [NA to NA] — not performed due to insufficient sera | 11 [4 to 21] | NA [NA to NA] — not performed due to insufficient sera | NA [NA to NA] — not performed due to insufficient sera | 22 [13 to 34]
  antiHBVtiter≥1.0 IU/mL-1m post (65,na,66,na,na,67) | 85 [74 to 92] | NA [NA to NA] — not performed due to insufficient sera | 92 [83 to 97] | NA [NA to NA] — not performed due to insufficient sera | NA [NA to NA] — not performed due to insufficient sera | 97 [90 to 100]

19. Secondary Outcome: ELISA GMT Concentrations for Routine Vaccines (Hib, Diphtheria, Tetanus, Hepatitis B) When Given Concomitantly With Novartis MenACWY Ad+ or Novartis MenACWY Ad- Conjugate Vaccines for Hib, Diphtheria, Tetanus, Hepatitis B
Description: To assess the Enzyme-linked immunosorbent assay (ELISA) GMT of Hib, Diphtheria, Tetanus, Hepatitis B, administered Concomitantly with Novartis MenACWY Ad+ or MenACWY Ad-conjugate vaccines, at the baseline and 1 month after primary vaccination by groups.
Time Frame: Baseline and 1 month after the 2 or 3 dose primary vaccination series
Population: The analysis was performed on the MenACWY per-protocol (PP) "n" population after primary vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 70 | 77 | 70 | 73 | 72 | 73
titers
  Tetanus - baseline (n=69,71,70,67,69,72) | 0.32 [0.24 to 0.41] | 0.31 [0.24 to 0.4] | 0.23 [0.18 to 0.29] | 0.28 [0.22 to 0.37] | 0.25 [0.19 to 0.32] | 0.18 [0.14 to 0.23]
  Tetanus - 1 m after 1st vacc(n=69,71,70,67,69,72) | 0.7 [0.57 to 0.87] | 0.92 [0.75 to 1.13] | 1.4 [1.14 to 1.72] | 0.6 [0.48 to 0.73] | 0.97 [0.79 to 1.19] | 0.68 [0.55 to 0.83]
  Diphtheria - baseline (n=69,71,70,67,69,72) | 0.035 [0.026 to 0.047] | 0.04 [0.03 to 0.053] | 0.027 [0.02 to 0.035] | 0.031 [0.024 to 0.042] | 0.032 [0.024 to 0.042] | 0.016 [0.012 to 0.021]
  Diphtheria -1m after 1st vacc(n=69,71,70,67,69,72) | 1.02 [0.81 to 1.29] | 1.02 [0.82 to 1.28] | 1.72 [1.38 to 2.14] | 1.06 [0.84 to 1.32] | 0.98 [0.78 to 1.22] | 1.49 [1.19 to 1.87]
  Hib - baseline (n=70,77,69,73,72,73) | 0.078 [0.056 to 0.11] | 0.15 [0.11 to 0.21] | 0.11 [0.078 to 0.15] | 0.089 [0.063 to 0.12] | 0.15 [0.11 to 0.21] | 0.064 [0.045 to 0.09]
  Hib - 1 m after 1st vacc (n=70,77,69,73,72,73) | 4.63 [3.14 to 6.83] | 4.55 [3.08 to 6.72] | 4.53 [3.07 to 6.68] | 0.47 [0.32 to 0.7] | 5.67 [3.89 to 8.28] | 0.42 [0.28 to 0.63]
  Hepatitis B - baseline (n=65,na,66,na,na,67) | NA [NA to NA] — not performed due to insufficient sera | NA [NA to NA] — not performed due to insufficient sera | 5.9 [4.25 to 8.2] | 5.79 [4.15 to 8.09] | NA [NA to NA] — not performed due to insufficient sera | 4.21 [3.03 to 5.87]
  Hepatitis B-1m after 1st vacc(n=65,na,66,na,na,67) | NA [NA to NA] — not performed due to insufficient sera | NA [NA to NA] — not performed due to insufficient sera | 378 [258 to 554] | 69 [47 to 102] | NA [NA to NA] — not performed due to insufficient sera | 133 [90 to 195]

20. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:4 and ≥ 1:8 Against N. Meningitidis Serogroup C Following 2 Doses of MenACWY Ad+ or Ad- Conjugate Vaccine (Containing 5 μg of MenC Oligosaccharide) or 2 Doses of Menjugate (Containing 10 μg of MenC Oligosaccharide)
Description: The immunogenicity was measured as percentages of subjects with hSBA ≥ 1:4 and ≥ 1:8 and associated 95% CI, directed against N. Meningitidis serogroup C, at baseline and 1 month after second vaccination by groups.
Time Frame: Baseline and 1 month after second vaccination
Population: The analysis was performed on the MenACWY and Menjugate per-protocol (PP) "n" population after second vaccination.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | UKMenC (Menjugate at 2, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 40 | 77 | 74 | 79 | 85
percentages of subjects
  hSBA ≥1:4, baseline | 23 [11 to 38] | 13 [6 to 23] | 15 [8 to 25] | 20 [12 to 31] | 20 [12 to 30]
  hSBA ≥1:4, 1 month after second vaccination | 98 [87 to 100] | 84 [74 to 92] | 91 [81 to 96] | 86 [76 to 93] | 93 [85 to 97]
  hSBA ≥1:8, baseline | 10 [3 to 24] | 9 [4 to 18] | 15 [8 to 25] | 5 [1 to 12] | 11 [5 to 19]
  hSBA ≥1:8, 1 month after second vaccination | 98 [87 to 100] | 83 [73 to 91] | 85 [75 to 92] | 82 [72 to 90] | 89 [81 to 95]

21. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After 2 or 3 Dose Primary Vaccination Series With MenACWY Ad+ or MenACWY Ad-
Description: Safety and tolerability of Novartis MenACWY Ad+ and MenACWY Ad- conjugate vaccine when given in a 2 or 3 dose primary vaccination series concomitantly with licensed pediatric vaccines.
Time Frame: 7 days after each vaccination
Population: Analysis was done on safety dataset "n" population - subjects who received at least one study dose and had Post baseline safety data.
Measure: Number; unit: subjects
Arm/Group | UK234+ (MenACWY Ad+ at 2, 3, 4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | UKMenC (Menjugate at 2, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m) | CA24+ (MenACWY Ad+ at 2, 4 m) | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m)
Number analyzed (Participants) | 90 | 90 | 45 | 98 | 98 | 90 | 90
subjects
  Tenderness | 40 | 31 | 18 | 46 | 32 | 41 | 35
  Erythema | 69 | 64 | 34 | 73 | 67 | 78 | 66
  Induration | 21 | 24 | 12 | 36 | 18 | 40 | 24
  Eating habit Change | 28 | 25 | 9 | 35 | 27 | 21 | 20
  Sleepiness | 56 | 49 | 25 | 64 | 62 | 45 | 52
  Persistent Crying | 7 | 7 | 6 | 15 | 4 | 5 | 4
  Irritability | 63 | 71 | 31 | 80 | 70 | 61 | 73
  Vomiting | 19 | 26 | 9 | 23 | 15 | 14 | 11
  Diarrhea | 29 | 27 | 12 | 30 | 22 | 18 | 16
  Fever (≥38°C) | 7 | 4 | 1 | 14 | 7 | 5 | 5
  Analgesics/Antipyretics | 43 | 35 | 18 | 61 | 46 | 36 | 45

22. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After MenACWY Ad+ and MenACWY Ad- Booster or Polysaccharide Challenge Administered at 12 Months of Age
Description: The safety profile of Novartis MenACWY Ad+ and MenACWY Ad- conjugate vaccines when given at 12 months of age.
Time Frame: 7 days after vaccination at 12 months of age
Population: Analysis was done on safety dataset "n" population.
Measure: Number; unit: subjects
Groups:
- UK234+ (MenACWY Ad+ at 2,3,4 m): Three doses of MenACWY conjugate vaccine with adjuvant were given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age. A fourth dose of MenACWY Ad+ was given at 12 months of age.
- CA246+ (MenACWY Ad+ at 2, 4, 6 m) - No Treatment: Three doses of MenACWY conjugate vaccine with adjuvant were given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was administered one dose of MMR (and Prevnar, if available) at 12 months of age.
- CA246+ (MenACWY Ad+ at 2, 4, 6 m) - PS; CA24+ (MenACWY Ad+ at 2, 4 m) - ACWY; CA24+ (MenACWY Ad+ at 2, 4 m) - PS: Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad+ vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- UK24- (MenACWY Ad- at 2, 4 m): Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad- vaccine was given at 12 months of age.
- CA24- (MenACWY Ad- at 2, 4 m) - ACWY: Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad- vaccine or one reduced dose (one fifth) of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- CA24- (MenACWY Ad- at 2, 4 m) - PS: Two doses of MenACWY conjugate vaccine with adjuvant were given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.
  One dose of MenACWY Ad- vaccine or one reduced dose of MenACWY PS vaccine was given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK234+ (MenACWY Ad+ at 2,3,4 m) | UK24+ (MenACWY Ad+ at 2, 4 m) | UKMenC (Menjugate at 2, 4 m) | CA246+ (MenACWY Ad+ at 2, 4, 6 m) - No Treatment | CA246+ (MenACWY Ad+ at 2, 4, 6 m) - PS | CA24+ (MenACWY Ad+ at 2, 4 m) - ACWY | CA24+ (MenACWY Ad+ at 2, 4 m) - PS | UK24- (MenACWY Ad- at 2, 4 m) | CA24- (MenACWY Ad- at 2, 4 m) - ACWY | CA24- (MenACWY Ad- at 2, 4 m) - PS
Number analyzed (Participants) | 90 | 90 | 45 | 48 | 48 | 47 | 48 | 90 | 44 | 43
subjects
  Tenderness | 7 | 11 | 10 | 0 | 10 | 7 | 10 | 10 | 7 | 12
  Erythema | 62 | 58 | 36 | 0 | 21 | 27 | 30 | 66 | 21 | 26
  Induration | 21 | 32 | 18 | 0 | 12 | 9 | 9 | 36 | 10 | 15
  Eating habit change | 11 | 16 | 5 | 10 | 12 | 6 | 10 | 13 | 10 | 8
  Sleepiness | 11 | 14 | 9 | 10 | 8 | 7 | 13 | 16 | 9 | 7
  Persistent crying | 0 | 4 | 3 | 3 | 3 | 0 | 2 | 4 | 5 | 0
  Irritability | 26 | 32 | 20 | 24 | 23 | 19 | 24 | 28 | 17 | 20
  Vomiting | 4 | 6 | 4 | 2 | 7 | 0 | 4 | 8 | 5 | 4
  Diarrhea | 9 | 9 | 4 | 4 | 7 | 6 | 5 | 9 | 3 | 4
  Fever (≥38°C) | 3 | 7 | 2 | 3 | 6 | 1 | 8 | 14 | 4 | 1
  Analgesics/Antipyretics | 14 | 21 | 12 | 13 | 15 | 8 | 17 | 22 | 14 | 11

ADVERSE EVENTS:
Time Frame: All solicited adverse events (AEs) were collected upto Day 7 after each vaccination. All SAEs and unsolicited AEs were collected throughout the study (22 months in total).
Description: Information on all AEs was to be collected for 7 days following each vaccination, after which information on only SAEs and AEs necessitating a physician's visit and/or resulting in premature withdrawal of subjects from the study was collected until the next study visit and recorded by study personnel.
Groups:
- UK234+ (MenACWY Ad+ at 2,3,4 m): Three doses of MenACWY Ad+ vaccine were to be given at 1-month intervals concomitantly with DTaPHibIPV at 2, 3, and 4 months of age. A fourth dose of MenACWY Ad+ was to be given at 12 months of age.
- UK24+ (MenACWY Ad+ at 2,4 m): Two doses of MenACWY Ad+ vaccine were to be given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad+ vaccine was to be given at 12 months of age.
- UKMenC (Menjugate at 2,4m): Two doses of Menjugate® were to be given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. One dose of MenACWY Ad+ vaccine was to be given at 12 months of age.
- CA246+ (MenACWY Ad+ at 2,4,6m): Three doses of MenACWY Ad+ vaccine were to be given at 2-month intervals concomitantly with DTaPHibIPV, HBV, and Prevnar® at 2, 4, and 6 months of age (Prevnar at 6 months was optional and was given if available). One subgroup of subjects was to be given a reduced dose of MenACWY PS vaccine concomitantly with MMR (and Prevnar, if available) at 12 months of age. Another subgroup was to be administered one dose of MMR (and Prevnar, if available) at 12 months of age.
- CA24+ (MenACWY Ad+ at 2,4m): Two doses of MenACWY Ad+ vaccine were to be given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar at 2 and 4 months of age.One dose of MenACWY Ad+ vaccine or one reduced dose (one fifth) of MenACWY PS vaccine was to be given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
- UK24- (MenACWY Ad- at 2,4m): Two doses of MenACWY Ad- vaccine were to be given at a 2-month interval concomitantly with DTaPHibIPV at 2 and 4 months of age. A third dose of MenACWY Ad- vaccine was to be given at 12 months of age.
- CA24- (MenACWY Ad- at 2,4m): Two doses of MenACWY Ad- vaccine were to be given at a 2-month interval concomitantly with DTaPHibIPV, HBV, and Prevnar® at 2 and 4 months of age.One dose of MenACWY Ad- vaccine or one reduced dose (one fifth) of MenACWY PS vaccine was to be given concomitantly with MMR (and Prevnar, if available) at 12 months of age.
Arm/Group | UK234+ (MenACWY Ad+ at 2,3,4 m) | UK24+ (MenACWY Ad+ at 2,4 m) | UKMenC (Menjugate at 2,4m) | CA246+ (MenACWY Ad+ at 2,4,6m) | CA24+ (MenACWY Ad+ at 2,4m) | UK24- (MenACWY Ad- at 2,4m) | CA24- (MenACWY Ad- at 2,4m)
Serious Adverse Events (participants affected / at risk) | 20/90 | 17/90 | 6/45 | 9/98 | 4/98 | 10/90 | 7/90
Other Adverse Events (participants affected / at risk) | 90/90 | 89/90 | 45/45 | 97/98 | 97/98 | 90/90 | 89/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UK234+ (MenACWY Ad+ at 2,3,4 m) (N=90) | UK24+ (MenACWY Ad+ at 2,4 m) (N=90) | UKMenC (Menjugate at 2,4m) (N=45) | CA246+ (MenACWY Ad+ at 2,4,6m) (N=98) | CA24+ (MenACWY Ad+ at 2,4m) (N=98) | UK24- (MenACWY Ad- at 2,4m) (N=90) | CA24- (MenACWY Ad- at 2,4m) (N=90)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
CONGENITAL MEGACOLON (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOSPADIAS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
PLAGIOCEPHALY (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
CYST (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEVELOPMENTAL DELAY (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
FOOD ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BRONCHIOLITIS (Infections and infestations) | 4 | 3 | 1 | 2 | 1 | 2 | 2
CROUP INFECTIOUS (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
INFECTED CYST (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
SALMONELLOSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VARICELLA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 4 | 2 | 1 | 1 | 0 | 0 | 0
VIRAL RASH (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
BURNS FIRST DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
FEBRILE CONVULSION (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACROCHORDON EXCISION (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
CIRCUMCISION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYDROCELE OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 | 0 | 0 | 2 | 0 | 0 | 0
TENDON SHEATH INCISION (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UK234+ (MenACWY Ad+ at 2,3,4 m) (N=90) | UK24+ (MenACWY Ad+ at 2,4 m) (N=90) | UKMenC (Menjugate at 2,4m) (N=45) | CA246+ (MenACWY Ad+ at 2,4,6m) (N=98) | CA24+ (MenACWY Ad+ at 2,4m) (N=98) | UK24- (MenACWY Ad- at 2,4m) (N=90) | CA24- (MenACWY Ad- at 2,4m) (N=90)
CONJUNCTIVITIS (Eye disorders) | 3 | 9 | 3 | 3 | 1 | 12 | 1
CONSTIPATION (Gastrointestinal disorders) | 7 | 1 | 2 | 8 | 6 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 41 | 40 | 18 | 37 | 34 | 36 | 25
VOMITING (Gastrointestinal disorders) | 24 | 37 | 13 | 29 | 23 | 28 | 20
CRYING (General disorders) | 7 | 11 | 8 | 19 | 8 | 14 | 9
INJECTION SITE ERYTHEMA (General disorders) | 79 | 79 | 40 | 73 | 78 | 84 | 68
INJECTION SITE INDURATION (General disorders) | 39 | 43 | 25 | 42 | 25 | 59 | 36
INJECTION SITE PAIN (General disorders) | 42 | 39 | 23 | 50 | 41 | 45 | 45
IRRITABILITY (General disorders) | 69 | 82 | 39 | 85 | 85 | 77 | 82
PYREXIA (General disorders) | 11 | 13 | 3 | 30 | 22 | 19 | 21
BRONCHIOLITIS (Infections and infestations) | 8 | 4 | 1 | 3 | 5 | 3 | 0
CROUP INFECTIOUS (Infections and infestations) | 1 | 0 | 0 | 3 | 5 | 1 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 8 | 0 | 2 | 0 | 9 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 13 | 14 | 0 | 14
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 2 | 5 | 1 | 0
OTITIS MEDIA (Infections and infestations) | 6 | 7 | 1 | 9 | 7 | 12 | 4
RHINITIS (Infections and infestations) | 30 | 34 | 15 | 2 | 0 | 39 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 10 | 8 | 21 | 25 | 3 | 20
VIRAL INFECTION (Infections and infestations) | 6 | 7 | 1 | 0 | 1 | 4 | 0
SOMNOLENCE (Nervous system disorders) | 58 | 57 | 29 | 68 | 70 | 57 | 63
EATING DISORDER (Psychiatric disorders) | 34 | 42 | 17 | 45 | 42 | 37 | 38
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 9 | 3 | 6 | 16 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 6 | 0 | 4
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5 | 2 | 0 | 3
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 6 | 3 | 1 | 6 | 7 | 2 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 4 | 1 | 5 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 8 | 13 | 5 | 15 | 8 | 8 | 7
RASH (Skin and subcutaneous tissue disorders) | 3 | 4 | 3 | 5 | 3 | 2 | 8
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigators from publishing. Any publications from a single site are postponed until the publication of the pool data (i.e., data from all sites) in the clinical trial.